CLINICAL TRIAL: NCT00984204
Title: Clinical Evaluation of Therapy™ Cool Path™ Duo Cardiac Ablation System for the Treatment of Typical Atrial Flutter (AFL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90030638
Record Dates: First submitted 2009-09-22; First posted 2009-09-25 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Typical Atrial Flutter
Keywords: cavo-tricuspid dependent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: Therapy Cool Path Duo

INTERVENTIONS:
Device: Therapy Cool Path Duo — All patients will be treated with Therapy Cool Path Duo Ablation System for the treatment of typical atrial flutter.

SUMMARY:
The purpose of this study is to demonstrate that ablation with the Therapy™ Cool Path™ Duo cardiac ablation system can eliminate typical atrial flutter and that its use does not result in an unacceptable risk of serious adverse events (SAE's).

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized study (historical data as control) for the evaluating the safety and efficacy of Therapy TM Cool PathTM

Duo Ablation System for the treatment of typical atrial flutter (Cavo-triscupid isthmus dependent)

ELIGIBILITY:
Inclusion Criteria:

* A signed written Informed Consent
* Presence of typical atrial flutter (cavotricuspid isthmus dependent)
* If subjects are receiving antiarrhythmic drug therapy (Class I or Class III AAD)for an arrhythmia other than typical atrial flutter, then the subject needs to be controlled on their medication for at least 3 months. If the subject had typical atrial flutter before starting the AAD(s) (Class I or Class III) and then subsequently had another arrhythmia (i.e. atrial fibrillation), then the 3 month AAD criteria will not apply.
* One documented occurrence of the study arrhythmia documented by ECG, Holter, telemetry strip, or transtelephonic monitor within the past 6 months
* In good physical health
* 18 years of age or older
* Agree to comply with follow-up visits and evaluation

Exclusion Criteria:

* Prior typical atrial flutter ablation treatment
* Pregnancy
* Atypical flutter or scar flutter(non-isthmus dependent)
* Significant coronary heart disease or heart failure; that is unstable angina pectoris and/or uncontrolled congestive heart failure (NYHA Class III or IV) at the time of enrollment
* A recent myocardial infarction within 3 months of the intended procedure date
* Permanent coronary sinus pacing lead
* Tricuspid valvular disease requiring surgery and/or a prosthetic tricuspid heart valve (i.e. significant)
* Evidence of intracardiac thrombus or a history of clotting disorders
* Participation in another investigational study
* Cardiac surgery within 1 month of the intended procedure date
* Allergy or contraindication to Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - Regional Cardiology Associates, Sacramento, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Moses Cone Hospital, Greensboro, North Carolina
  - Ohio State Medical, Columbus, Ohio
  - Cardiovascular Associates of Cleveland, Mayfield Heights, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Main Line Health Center/Lankenau, Wynnewood, Pennsylvania
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Virginia Hospital Center, Arlington, Virginia
  - University of Virginia Medical Center, Charlottesville, Virginia
- Canada (2):
  - Victoria Cardiac Arrhythmia Trials, Inc., Victoria, British Columbia
  - Institut de Cardiologie de Quebec, Québec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 188
Completed | 173 (Seven subjects of the ten "Lack of efficacy" were acute failures that had no block after 30 min)
Not Completed | 15
Not completed — Death | 1
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 10

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.47 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 160
Region of Enrollment [Number; unit: participants]
  United States | 162
  Canada | 26

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety- Incidence of Intra Procedural Serious Cardiac Adverse Events Occuring Within 7 Days of Post-procedure, Regardless of Whether a Determination Can be Made Regarding Device Relatedness.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 188
participants | 12 [3.34 to 10.88]

2. Primary Outcome: Primary Efficacy- Bidirectional Block in the Cavo-tricuspid Isthmus and Non-inducibility of Typical Atrial Flutter at Least 30 Minutes Following the Last RF Ablation With the Cool Path Duo Ablation Catheter System is Obtained.
Time Frame: 30 mins
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 188
participants | 181 [93.57 to 98.98]

3. Secondary Outcome: Secondary Efficacy- Freedom From Recurrence of Typical Atrial Flutter up to 3 Months Post Procedure
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 188
participants | 173 [91.24 to 97.83]

ADVERSE EVENTS:
Time Frame: Composite SAEs within 7 days
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 12/188
Other Adverse Events (participants affected / at risk) | 23/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=188)
Cardiac Arrhythmia (Cardiac disorders) | 3
Congestive Heart Failure (Cardiac disorders) | 2
Syncope (Nervous system disorders) | 1
Pericarditis (Injury, poisoning and procedural complications) | 1
Coronary Artery Disease (Vascular disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=188)
Cardiac Arrhthymia (Cardiac disorders) | 20
Palpitations (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No